CLINICAL TRIAL: NCT03916354
Title: Clinical Study of the Effect of Gestational Weight Gain on Composition of Gut Microbiome
Brief Title: Maternal Gestational Weight Gain and Microbiota of Maternal and Infant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liangkun Ma, Deputy professor of obstetrics and gynecology, Peking Union Medical College Hospital
Other Study IDs: HS-1875
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Pregnancy; Gestational Weight Gain; Microbiota
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- appropriate GWG group: 2009 IOM criteria recommended an appropriate range of weight gain during pregnancy and during each pregnant trimester according to BMI. The participants whose GWG value is in the recommended normal range is in this group.
- excess GWG group: 2009 IOM criteria recommended an appropriate range of weight gain during pregnancy and during each pregnant trimester according to BMI. The participants whose GWG value is over the upper limit of the recommended normal range is in this group.
- insufficient GWG group: 2009 IOM criteria recommended an appropriate range of weight gain during pregnancy and during each pregnant trimester according to BMI. The participants whose GWG value is below the lower limit of the recommended normal range is in this group.

SUMMARY:
A prospective, multicenter, observational cohort study including about 550 mother-infant pairs in Beijing will be conducted to evaluate the association between mothers' gestational weight gain and the gut microbiota of them and their infants.

DETAILED DESCRIPTION:
Purpose To evaluate whether mothers' gestational weight gain is associated with differences in maternal and their infants gut microbiota characteristics.

Methods and analysis This is a prospective, multicenter, observational cohort study including about 550 mother-infant pairs from PUMCH and other 3 hospitals in Beijing. After signing consent form, every participant will bring home a weighting scale for checking and record the weight every week from they enrolled to a year postpartum. The blood samples, fecal samples, vaginal swabs and oral swabs of the mothers will be collected at first, second, third trimester and postpartum 42 days. The infants' fecal samples will be collected at 0~3, 14, 42 days and 3, 6, 9, 12 months after born. Questionnaire for mothers (diet, exercise, antibiotic and probiotic usage, oral hygiene habits etc.) and their infants (delivery mode, feeding pattern, antibiotic and probiotic usage etc.), as well as the medical records will be collected along with the sample collecting. Bio-specimen will be tested by 16S rRNA gene sequencing. Logistical regression and covariance analysis will be used to determine the relationships between the demographic data, gestational weight gain and microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Ensure a regular prenatal check in the clinical centers.
* 20-45 years old.
* 8-13 gestational weeks.
* Singleton.
* Fully understand and voluntarily sign the informed consent.

Exclusion Criteria:

* IUI or IVF-ET pregnancy.
* Smoking or drinking.
* Antibiotics exposure within a month.
* With metabolic syndrome, hypertension, diabetes or dyslipidemia before pregnancy.
* With digestive disease, uncontrolled thyroid disease.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only pregnancies meet the criteria will be included in this study
Study Population: About 550 pregnant women meeting the conditions will be recruited from April 2019 to December 2019 during their routine antenatal caer at the first visit.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
maternal gut microbiota, vaginal microbiota, oral microbiota | From enrollment to 42 days postpartum
  The outcome will be measured at first, second and third trimester, as well as 42 days postpartum.
gut microbiota infants | From delivery to 1 year postpartum.
  The outcome will be measured at seven specific time points after the babies delivered.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Medical Univercity College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All data put together will only be shared by PUMCH and the company, but the article signature will be decided according contribution of the sub-centers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After finish the 2-year follow-up and the article of the whole data is received.
Access Criteria: Each sub-center complete their own task of enrollment and follow-up.

DOCUMENTS (1):
  • Informed Consent Form (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03916354/ICF_000.pdf